CLINICAL TRIAL: NCT01257191
Title: Cellular Inflammation Characterization of Nasal Challenges With Fine and Ultrafine Particles
Brief Title: A Study to Compare the Effects of Different Sized Particles on Cells in the Nose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Maria I. Garcia-Lloret, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: DAIT AADCRC-UCLA-02
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Hypersensitivity, Immediate; Atopic Hypersensitivity
Keywords: Vehicle Emissions; Diesel Exhaust
MeSH Terms: conditions — Hypersensitivity, Immediate | interventions — Soot; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Carbon Black (Experimental)
  Interventions: Drug: Carbon Black
- Diesel Exhaust Particles (Experimental)
  Interventions: Drug: Diesel Exhaust Particles
- Fine Concentrated Ambient Particles (Experimental)
  Interventions: Drug: Fine Concentrated Ambient Particles
- Ultrafine Concentrated Ambient Particles (Experimental)
  Interventions: Drug: Ultrafine Concentrated Ambient Particles
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Carbon Black — source: commercial
  Arms: Carbon Black
Drug: Diesel Exhaust Particles — source: diesel engine
  Arms: Diesel Exhaust Particles
Drug: Fine Concentrated Ambient Particles — source: concentrated ambient air
  Arms: Fine Concentrated Ambient Particles
Drug: Ultrafine Concentrated Ambient Particles — source: concentrated ambient air
  Arms: Ultrafine Concentrated Ambient Particles
Drug: Saline — Saline solution
  Arms: Placebo

SUMMARY:
The goal of this study is to see how the type and size of particles found in air pollution affects inflammation in the nose in people who are skin test positive to at least one allergen. It has been observed that pollution makes allergies worse. It has also been suggested that very small particles may affect allergies more than larger particles.

DETAILED DESCRIPTION:
Cough, bronchitis, asthma, and chronic obstructive pulmonary disease are all associated with elevated pollution particle levels. Researchers believe that particulate pollutants can exacerbate allergy and inflammation and affect asthma and allergy prevalence. In an urban setting such as the Los Angeles Basin, particles generated by vehicular traffic are thought to be important risk factors. Recently, the Environmental Health Centre of Southern California confirmed that there is a strong association between traffic near homes and schools and development of asthma. This study will help researchers describe the effects of various size pollution particles in causing inflammation in the nose.

There will be a total of 20 study visits. The study procedures include physical exams, symptom score for nose, nose washes and nose challenges with particulate matter. The particulates will be given in a random order and include the following: saline (sterile salt water), inert carbon particles (Carbon Black), diesel exhaust particles (DEP), small (fine) particles or very small (ultrafine) particles. These last two (fine and ultrafine) particles are obtained from concentrated normal Los Angeles air. The particulate will be sprayed into the nose with a standard nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Previously determined high inflammatory responders to Diesel Exhaust Particles
* Previously determined atopy as demonstrated by allergy skin testing
* Asymptomatic on day of challenge.

Exclusion Criteria:

* History of lung problems (including asthma), bleeding, neuromuscular, liver, kidney or heart disorders.
* History of anaphylaxis.
* Recent upper respiratory infection (less than 4 weeks prior to study) or other active infection.
* Active smoker or smoker in the past 2 years.
* Treatment with topical nasal steroids (< 1 month), systemic steroids (<1 month), oral antihistamines (< 1 week) prior to any nasal challenge.
* Use of leukotriene receptor antagonist (< 1 month ) prior to any nasal challenge
* Intranasal antihistamine or cromolyn use < 1 week prior to any nasal challenge .
* History of treatment with allergy immunotherapy.
* Inability to perform nasal lavage.
* Inability to give written informed consent
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The number of inflammatory cells in nasal lavage samples after exposure to 4 different types of particles | 6 and 24 hours after nasal challenge

SECONDARY OUTCOMES:
Differential cell count in nasal lavages | 6 and 24 hours post challenge
IL-8 in nasal lavages | 6 and 24 hours post challenge
TNFα in nasal lavages | 6 and 24 hours post challenge
RANTES in nasal lavages | 6 and 24 hours post challenge
MCP-1 in nasal lavages | 6 and 24 hours post challenge
MIP-1α in nasal lavages | 6 and 24 hours post challenge
GM-CSF in nasal lavages | 6 and 24 hours post challenge
Nitrite in nasal lavages | 6 and 24 hours post challenge
Induced ROS generation (presence of intracellular thiol, 8-Isoprostane, and hydrogen peroxide) in nasal lavage cells | 6 and 24 hours post challenge
Phase II enzymes (HO-1, GSTP1, NQO1 and GSTM1) in nasal lavage | 6 and 24 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: Maria G Lloret, MD, Study Chair — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov